CLINICAL TRIAL: NCT03986125
Title: Emotional Awareness and Expression Therapy and Mindfulness Meditation Training for College Students With Anxiety and Somatic Symptoms: A Randomized Controlled Trial
Brief Title: Student Anxiety & Stress Study
Acronym: SASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Distinguished Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1904002172
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Anxiety; Somatic Symptom Disorder
Keywords: college students; anxiety; somatic symptoms
MeSH Terms: conditions — Anxiety Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Masking Description: Prior to randomization all parties will be blinded to experimental condition. Post treatment and follow up assessments will be conducted by a blinded research assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Awareness & Expression Therapy (Experimental): Participants will attend three individual sessions focused on becoming aware of and expressing avoided or conflicted emotions.
  Interventions: Behavioral: Emotional Awareness & Expression Therapy
- Mindfulness Meditation Training (Experimental): Participants will attend three individual sessions focused on increasing equanimity and compassion and reducing self-judgement.
  Interventions: Behavioral: Mindfulness Meditation Training
- Wait-List Control (No Intervention): Participants will receive the intervention of their choice following assessment at four and eight weeks after randomization.

INTERVENTIONS:
Behavioral: Emotional Awareness & Expression Therapy — emotion-focused
  Arms: Emotional Awareness & Expression Therapy
Behavioral: Mindfulness Meditation Training — meditation training and practice
  Arms: Mindfulness Meditation Training

SUMMARY:
The present study is a randomized clinical trial of an emotional awareness and expression intervention (EAET) and a mindfulness meditation intervention (MMT) for Wayne State University students with anxiety and somatic symptoms. Each of these treatments will be compared to a wait list control condition and to one another to evaluate how well the treatments improve physical and psychological symptoms, stress, and interpersonal functioning of 120 Wayne State University students at 4-week and 8-weeks post-randomization. This research is intended to provide an evidence-based approach to working with emotions to improve both anxiety and somatic symptoms in young adults and will illuminate how EAET compares to the commonly used mindfulness training. It is hypothesized that both active interventions will be superior to no treatment, and differences between the two treatments will be explored.

DETAILED DESCRIPTION:
Anxiety is an increasingly common condition among college students and is often accompanied by somatic symptoms. These conditions impair students' social, psychological, and academic functioning and outcomes. Although students are utilizing campus and community mental health centers at increasing rates, these resources are strained. The present study aims to test the efficacy of two brief treatment options for students.

Integrating techniques from several emotion-focused therapies, the investigators have developed and tested an intervention encouraging the awareness and expression of habitually suppressed or avoided emotions. This Emotional Awareness and Expression Therapy (EAET) has been evaluated with various patient populations including fibromyalgia, irritable bowel syndrome, chronic pelvic pain, and medically unexplained symptoms. Results of these trials suggest that the intervention is efficacious in improving physical and psychological well-being, and is equal to or superior to other psychological interventions for somatic conditions. The present study seeks to advance the EAET literature by evaluating the efficacy of the intervention for a broader population and by employing a strong and conceptually different comparison condition: mindfulness meditation training.

ELIGIBILITY:
Inclusion Criteria: university student, reporting at least moderate levels of anxiety (GAD-7) and somatic symptoms (PHQ-15) -

Exclusion Criteria: psychosis, lack of fluency with spoken and written English language

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Scale-7 | change from baseline to four and eight weeks after baseline
  symptoms of anxiety
Patient Health Questionnaire-15 | change from baseline to four and eight weeks after baseline
  The 15-item measure asks patients how much they have been bothered by various somatic symptoms such as headaches, back pain, and digestive distress during the previous 2 weeks, with answers ranging from 0 (not at all) to 2 (a lot). Items are summed to generate a total score with higher scores indicating greater distress regarding somatic symptoms.

SECONDARY OUTCOMES:
Brief Symptom Inventory | change from baseline to four and eight weeks after baseline
  psychological symptoms
Patient Global Impression of Change | four and eight weeks after baseline
  change in health status since the start of the study
Perceived Stress Scale | change from baseline to four and eight weeks after baseline
  The 14-item measure asks patients how often they had experienced thoughts and feelings such as lack of control and difficulty coping during the previous 2 weeks, with answers ranging from 0 (never) to 4 (very often). Items are summed to generate a total score with higher scores indicating higher levels of perceived stress.
Satisfaction With Life Scale | change from baseline to four and eight weeks after baseline
  The 5-item measure asks patients the degree to which they agree with statements such as "In most ways my life is close to my ideal", with answers ranging from 1 (strongly disagree) to 7 (strongly agree). Items are summed to create a total score with higher scores indicating a greater degree of satisfaction with life.

OTHER OUTCOMES:
Emotional Approach Coping Scale | change from baseline to four and eight weeks after baseline
  emotional approach coping
Emotional Expressivity Scale | change from baseline to four and eight weeks after baseline
  Measures the extent to which patients outwardly display emotion. The 17-item measure asks patients the degree to which items such as "I display my emotions to other people" describe them on a scale from 1 (never) to 6 (always). Scores are summed to generate a total score with higher scores indicating greater emotional expressiveness.
Cognitive and Affective Mindfulness Scale-Revised | change from baseline to four and eight weeks after baseline
  The 12-item measure asks patients to rate the degree to which statements indicating four components of mindfulness (attention, focus on the present, awareness, and acceptance) apply to them, on a scale ranging from 1 (rarely/not at all) to 4 (almost always). Items are summed to generate a total score with higher scores indicating greater mindfulness.
Acceptance and Action Questionnaire | change from baseline to four and eight weeks after baseline
  ). The 9-item measure assesses avoidance of private experiences such as emotions, thoughts, and memories as well as the ability to take action under adverse circumstances. It asks patients to indicate how true each statement is of themselves on a scale ranging from 1 (never true) to 7 (always true). Items are summed and higher scores indicate greater levels of psychological inflexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No